CLINICAL TRIAL: NCT01022918
Title: Evaluation of the Irinotecan/Bevacizumab Association as Neo-adjuvant and Adjuvant Treatment of Chemoradiation With Temozolomide for Naive Unresectable Glioblastoma. Phase II Randomized Study With Comparison to Chemoradiation With Temozolomide
Brief Title: Evaluation of the Irinotecan/Bevacizumab Association for Naive Unresectable Glioblastoma
Acronym: TemAvIr
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Collaborators: National Cancer Institute, France (Other Government); Association de Neuro-Oncologues d'Expression Francaise (Other); UNICANCER (Other); Hoffmann-La Roche (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TemAvIr
Record Dates: First submitted 2009-11-26; First posted 2009-12-01 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Naive Unresectable Glioblastoma
Keywords: unresectable glioblastoma
MeSH Terms: interventions — Bevacizumab; Irinotecan; Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab/Irinoecan (Experimental): Neoadjuvant Treatment Patient will receive bevacizumab 10mg/kg plus irinotecan 125mg/m² 4 times every two weeks.
  Radiochemotherapy Then they will receive conformational radiotherapy for 6 weeks (30 Gy, 2Gy/fractions) associated with Temodal ( 75mg/m²/day) from first day up to the end of radiotherapy and 4 injections of Avastin (15mg/kg Day 1, day 15, day 29 and day 43).
  Adjuvant treatment:
  Patients will receive bevacizumab 15mg/kg plus irinotecan 125mg/m² 12 times every two weeks.
  Interventions: Drug: Avastin + Campto / radiotherapy + Temodal + Avastin (4 cures)
- Stupp (Active Comparator): patient will receive 6 weeks chemotherapy treatment associating conformational 30 Gy (2Gy/ fraction)and Temodal(75mg/m²/day, followed by 6 months adjuvant therapy consisting in 5 days every 28 days of Temodal (150-200mg/m².
  Interventions: Drug: Temodal/radiotherapy

INTERVENTIONS:
Drug: Avastin + Campto / radiotherapy + Temodal + Avastin (4 cures)
  Arms: Bevacizumab/Irinoecan
Drug: Temodal/radiotherapy
  Arms: Stupp

SUMMARY:
Treatment of glioblastoma (GBM) is based on surgery when possible, and chemoradiation with temozolomide, which became a standard since the EORTC study (Stupp, 2005). However, the prognosis of unresectable GBM remains poor despite chemoradiation with an estimated 10 month median survival, in the range of the comparable patients in the RPA class V from the EORTC study (Miramanoff, 2006).

Vredenburgh et al. from the Duke University (Durham, NC) reported at ASCO 2006 (fully published in J Clin Oncol, 2007) a 57 % unexpected response rate using a bevacizumab/irinotecan schedule in patients with relapsed GBM or grade 3 astrocytomas. This unusual high response rate, sometimes with major and sustained responses, was confirmed by a cooperative french study of ANOCEF (Guiu et al., 2008). Such a major improvement of treatment effectiveness lead ANOCEF, which federates most of the active neuro-oncology teams in France, to propose a neo-adjuvant and adjuvant bevacizumab-based chemotherapy framing a standard temozolomide-based chemoradiation with the aim to improve the prognosis of unresectable GBM.

The bevacizumab/temozolomide combination as neo-adjuvant is presently being evaluated by the Duke University. We believe that an ambitious comparison of the bevacizumab/irinotecan-schedule with the ''standard'' temozolomide-based chemoradiation is a fascinating challenge to improve the treatment of this awful disease.

The ANOCEF proposal '' Evaluation of the irinotecan/bevacizumab association as neo-adjuvant and adjuvant treatment of chemoradiation with temozolomide for naive unresectable glioblastoma. Phase II randomized study with comparison to chemoradiation with temozolomide'' has been successfully granted by INCA (Institut National du Fancer, France) through its research program ( PHRC : Programme Hospitalier de Recherche Clinique). Implementation of this program is now starting .

ELIGIBILITY:
Inclusion Criteria:

All the eligibility criteria must be met before registration :

* delay upper or equal to 14 days from stereotaxic biopsy and 28 days from surgical biopsy
* Histopathologically proven diagnosis of glioblastoma (WHO grade IV astrocytoma)
* Patient belonging to the RPA V class or associated
* only supratentorial glioblastoma
* Diagnosis must be obtained by a stereotactic or surgical biopsy
* Age between 18 and 70
* A contrast-enhanced MRI must be performed within 28 days prior to study registration
* Total or partial surgical resection deemed as not possible by a neurosurgeon
* Karnofsky Index (KI) performance status over 50
* Life expectancy of at least 3 months
* A stable dose of corticosteroid for at least 7 days to control intracranial pressure and neurological symptoms
* Adequate blood function : absolute neutrophil count > 1.5 x 109/L, platelets count > 100 x 109/L platelets; hemoglobin > 10 g/dl after blood transfusion if required
* Adequate liver function: bilirubin < 1.5 ULN (upper limit of normal), ALT and AST < 2.5 ULN, Prothrombin rate > 75 %
* Adequate renal function: creatinine < 1.2 ULN; proteinuria test 0 or trace (or urine protein concentration < 1g/24h if proteinuria test is + or ++).
* Negative pregnancy test for women of childbearing potential and adequate contraception for men and women.
* systolic arterial blood pressure at rest ≤ 170 mmHg
* Patient must have been informed and must have signed the specific informed consent form.
* holder of a coverage by the health insurance

Exclusion Criteria:

* patient belonging to the RPA III or IV
* prior malignant tumor in the recent 5 years or concomitant malignancy
* prior anti-tumoral chemotherapy or radiotherapy
* prior gross resection of the brain tumor
* patient receiving gliadel
* cardiovascular contra-indications to bevacizumab : prior angina pectoris, prior myocardial infarction, prior brain stroke, even transient, distal severe arteriopathy, uncontrolled high blood pressure
* anticomitial drug p450 cytochrome inductors
* other substances inducing p450 cytochrome
* proteinuria ≥ 1g/L
* concurrent anticoagulant or platelet anti-aggregant treatment
* congenital haemorrhagic pathology (haemophilia, Willebrandt)
* sign of brain haemorrhage on the RMI initial exam
* non resolved infectious disease
* non controlled arterial hypertension (≥170 mmHg)
* intracranial high pressure not controlled by a stable dose of steroids for at least 7 days
* pregnancy or refusal of the contraception for women and men
* psychiatric, behavioural disorders or geographical situation precluding the administration or follow-up of the protocol (including claustrophobia)
* digestive haemorrhage and / or gastro-duodenal ulcer occurring in the last 3 months
* pregnant, nursing woman, or without contraception
* private individuals of freedom or under tutelage (including legal guardianship)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To determine the rate of non-progressive disease at 6 months after inclusion in each arms | after half of each arms has been completed at 6 months of treatment

SECONDARY OUTCOMES:
To determine if bevacizumab-based regimen increases the overall survival in comparison of the Stupp regimen | december 2011
To evaluate if any bevacizumab-based regimen increases the survival without neurologic degradation and the quality of life according to the QLC-C30 and the specific Brain Cancer Module QLQ-BN20 scales. | december 2011
To evaluate the tolerance of the bevacizumab-based regimens according to the NCI-CTCAE, version 3.0 scale. To record the rate of serious adverse events (mainly the theoretical risk of brain hemorrhage with bevacizumab) | december 2011

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Chauffert, Professor, Principal Investigator — Centre Hospitalier Universitaire, Amiens
Locations (1):
- Centre Georges François Leclerc, Dijon, Bourgogne-Franche-Comté, France

REFERENCES:
- [Derived] Chauffert B, Feuvret L, Bonnetain F, Taillandier L, Frappaz D, Taillia H, Schott R, Honnorat J, Fabbro M, Tennevet I, Ghiringhelli F, Guillamo JS, Durando X, Castera D, Frenay M, Campello C, Dalban C, Skrzypski J, Chinot O. Randomized phase II trial of irinotecan and bevacizumab as neo-adjuvant and adjuvant to temozolomide-based chemoradiation compared with temozolomide-chemoradiation for unresectable glioblastoma: final results of the TEMAVIR study from ANOCEFdagger. Ann Oncol. 2014 Jul;25(7):1442-1447. doi: 10.1093/annonc/mdu148. Epub 2014 Apr 9. PMID 24723487